CLINICAL TRIAL: NCT05901038
Title: Development of Artefact Removal and Physical Activity Algorithm for Continuous Activity Monitoring by Heart Rate Monitors in Cardiac Patients
Brief Title: Development of Artefact Removal and Physical Activity Algorithm
Acronym: ARTEPHYSICAL
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Universiteit Antwerpen (Other)
Responsible Party: Sponsor
Other Study IDs: ARTEPHYSICAL / EC 5241
Record Dates: First submitted 2023-05-02; First posted 2023-06-13 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-03

CONDITIONS: Exercise; Fitness Tracker; Heart Rate
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Cardiac patients (group 1): Patients with prior myocardial infarction, percutaneous coronary intervention (PCI), cardiac ablation or cardiac surgery, attending a reimbursed cardiac rehabilitation programme in the cardiology department of the UZA.
  Interventions: Device: Wearing heart rate monitors
- Coached sporters with 12-week training schedule (group 2): Sporters attending a sports cardiology consultation and following a 12-week training schedule at Sport Medical Centre Nottebohm.
  Interventions: Device: Wearing heart rate monitors
- Sporters without 12-week training schedule (group 3): Sporters attending a sport medical check-up at S.P.O.R.T.S. (i.e., a multidisciplinary centre of expertise within UZA), but without standardized 12-week training schedule.
  Interventions: Device: Wearing heart rate monitors

INTERVENTIONS:
Device: Wearing heart rate monitors — Participants will use 2 consumer wearable heart rate monitors: Polar H10 chest strap and Fitbit Inspire 2 fitness tracker.

SUMMARY:
This clinical trial will collect heart rate (HR) data with the Fitbit Inspire 2 fitness tracker and Polar H10 chest strap with the aim of:

* Goal 1. Optimising and validating our artefact removal procedure.
* Goal 2. Developing a physical activity (PA) algorithm to follow and quantify day-to-day PA based on HR measurements.

A pilot study will be conducted with a total of 46 cardiac patients (group 1), 46 coached sporters with 12-week training schedule (group 2) and 46 sporters without 12-week training schedule (group 3). The three groups all engage in controlled activities.

The participants' HR will be monitored continuously for an average period of 13 weeks using 2 HR monitors, i.e. the Fitbit Inspire 2 fitness tracker and the Polar H10 chest strap. They will wear the Fitbit device continuously for the whole monitoring period, while they will wear the Polar chest strap continuously for the first 24 hours and after that only during exercise.

To determine participants' exercise capacity (e.g. VO2max), cardiopulmonary exercise tests (CPETS) will be carried out. For group 1, 3 CPETS will take place during the CR programme: at the start, in the middle and at the end. For group 2 and group 3, 2 CPETS will be carried out at the start and the end of the study. The monitoring period with Fitbit and Polar will end at the last CPET.

All participants will record their daily efforts in an activity diary during the first week of study. Moreover, two questionnaires will be conducted at the end of the study to evaluates usability and experiences with the HR monitors.

DETAILED DESCRIPTION:
Sufficient physical activity (PA) is becoming more and more important in the prevention, onset and treatment of several cardiovascular diseases. Heart rate (HR) monitors are of interest to researchers and various healthcare providers because of their ability to use HR to indicate PA levels of individual cardiac patients in an objective, accurate and continuous way.

However, artefacts such as over- and underestimation may affect the accuracy of these HR monitors in daily living conditions of specific cardio populations. Moreover, reliable parameters and algorithms to objectively map, calculate and monitor PA are still lacking.

The research group has been able to improve the accuracy of HR monitors by detecting and correcting artefacts and is further exploring the technical possibilities of developing an artefact removal procedure, aiming for an improved and automatic way to continuously monitor HR in cardiac patients. However, more data is needed to optimise and validate the procedure. In addition, more HR data of controlled activities are needed because the investigators aim to develop an innovative PA algorithm that calculates a daily score to quantify PA levels based on HR measurements and focused on the prediction of VO2max data (i.e. the gold standard indicator for determining exercise capacity).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years,
2. Patients participating in the CR programme with a prior myocardial infarction without impairment of pump function, percutaneous coronary intervention (PCI), cardiac ablation or cardiac surgery, OR Sporters attending a sports cardiology consultation and following a 12-week training schedule at Sport Medical Centre Nottebohm, OR Sporters attending a sport medical check-up at S.P.O.R.T.S. who do not follow a 12-week training schedule,
3. Having a smartphone available,
4. Being capable of signing the informed consent.

Exclusion Criteria:

1. Patients with severe heart failure (NYHA III-IV),
2. Not able to speak and read Dutch or English,
3. Cognitive impaired (e.g. severe dementia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Groups are selected from different populations: patients participating in a cardiac rehabilitation programme at the UZA (group 1), sporters attending a sports cardiology consultation at Sport Medical Centre Nottebohm (group 2) or sporters attending a sports medical check-up at S.P.O.R.T.S. (i.e., a multidisciplinary centre of expertise within UZA, group 3).
Sampling Method: Non-Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2023-02-24 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
A physical activity algorithm with accompanying score | During the entire duration of the study, on average 13 weeks
  The primary outcome of this study is an algorithm and associated score that quantifies day-to-day physical activity.

SECONDARY OUTCOMES:
Validation artefact removal procedure | During the entire duration of the study, on average 13 weeks
  The accuracy, sensitivity and specificity of the artefact removal procedure will be evaluated.
Satisfaction heart rate monitors | At study completion, on average after 13 weeks
  We will evaluate how participants perceive wearing heart rate monitors for long periods of time using self-developed questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Hein Heidbuchel, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University Hospital Antwerp, Edegem, Antwerp, Belgium